CLINICAL TRIAL: NCT01672060
Title: A Scientific Evaluation of the Nurse-Family Partnership (NFP) Program in British Columbia
Brief Title: BC Healthy Connections Project
Acronym: BCHCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Collaborators: McMaster University (Other); Ministry of Health, British Columbia (Other Government); Ministry of Children and Family Development, British Columbia (Other); University of British Columbia (Other); University of Victoria (Other); Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Principal Investigator, Dr. Charlotte Waddell, University Professor, Simon Fraser University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010s0569
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Effectiveness of Nurse-Family Partnership (NFP) in BC

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nurse-Family Partnership (NFP) (Experimental)
  Interventions: Behavioral: Nurse-Family Partnership (NFP)
- Existing services (Active Comparator)
  Interventions: Behavioral: Existing services

INTERVENTIONS:
Behavioral: Nurse-Family Partnership (NFP) — Trained Public Health Nurses (PHNs) will deliver Nurse-Family Partnership (NFP) using specified pregnancy, infancy and toddler curricula. Following enrollment in the study, NFP PHNs will provide regular home visits to participants throughout the remainder of the participant's pregnancy, continuing through until the child's second birthday. In addition to offering standard care during each visit, PHNs will deliver NFP content using program materials relevant to the following domains: personal health, maternal role, environmental health, family and friends, life course development, and health and human services.
  Arms: Nurse-Family Partnership (NFP)
Behavioral: Existing services — Participants allocated to the comparison group will receive all the usual perinatal programs and services offered within their Health Authority, including primary care and specialist physician services covered under BC's public healthcare system. These services vary across the province but may include: standard primary healthcare services; public health programs including prenatal classes, pregnancy outreach and home visiting by nurses or paraprofessionals; and a variety of targeted and universal parenting and early child development programs.
  Arms: Existing services

SUMMARY:
Nurse-Family Partnership (NFP) is a primary prevention program that was developed by Dr. David Olds in the United States (US) with the goal of helping vulnerable young first-time mothers and their children. The program involves public health nurses (PHNs) visiting mothers in their homes, providing intensive supports starting in pregnancy and continuing until children reach their second birthday. Studies in the US have shown that NFP significantly reduces child maltreatment and child behaviour problems, while also improving children's early learning and mother's economic self-sufficiency. Economic studies have also shown that the program pays for itself over the long-term. However, NFP has never been tested in Canada. Due to major differences in our populations and in our public services, we do not know whether NFP will show the same benefits here. We therefore plan to conduct a scientific evaluation of NFP's effectiveness in British Columbia (BC), in close collaboration with the BC government and BC's Health Authorities. Using randomized-controlled trial methods, NFP's effectiveness will be specifically evaluated in comparison with existing perinatal services in BC regarding outcomes across three fundamental domains: 1) pregnancy and birth; 2) child health and development; and 3) maternal health and life course. Findings from this evaluation will be used to improve the NFP program - to better meet the needs of vulnerable young mothers and their children in BC.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 24 years or under
2. First Birth
3. Less than 27 weeks gestation
4. Competent to provide informed consent, including conversational competence in English
5. Experiencing socioeconomic disadvantage (must meet 5a or 5b):

5a. Aged 19 years or younger (eligible) 5b. Aged 20-24 (eligible if has TWO of the following):

* 5.1. Lone parent (is not married or living common-law, i.e., not living with the same person for more than one year)
* 5.2. Less than grade 12 (does not have BC's Dogwood certificate, General Education Development [GED] Credential or other diploma equivalent to grade 12; note that the Evergreen Certificate is not equivalent to grade 12)
* 5.3. Low income (based on answering "yes" to any ONE of the following)
* 5.3a. Do you receive income assistance (e.g., disability, social assistance, employment insurance, or BC Medical Services Plan Premium Assistance)?
* 5.3b. Do you find it very difficult to live on your total household income, particularly regarding food and rent?
* 5.3c. Do you live in a group home, shelter, or institutional facility (e.g., treatment center)?

Exclusion Criteria:

1. Planning to have the child adopted
2. Planning to leave the NFP catchment area (for three months or longer)

Max Age: 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 739 (Actual)
Dates: Start 2013-10-15 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Average number of childhood injuries | 2, 10, 18 and 24 months postpartum
  The average number of physician/health care provider encounters per child for injuries (intentional or unintentional), measured in community/outpatient, emergency room (ER) and hospital settings, from birth through 24 months postpartum

SECONDARY OUTCOMES:
Prenatal substance use | Baseline (before 28 weeks gestation), 34-36 weeks gestation
  Tobacco and alcohol use
Child development | 24 months postpartum
  Cognitive ability and language development
Child mental health | 24 months postpartum
  Behaviour problems
Maternal life course | 2, 10, 18 and 24 months postpartum
  Number of subsequent pregnancies by 24 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Waddell, MSc, MD, CCFP, FRCPC, Principal Investigator — Director, Children's Health Policy Centre, Faculty of Health Sciences, Simon Fraser University
Locations (1):
- Children's Health Policy Centre, Faculty of Health Sciences, Simon Fraser University, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Catherine NLA, MacMillan H, Jack S, Zheng Y, Xie H, Boyle M, Sheehan D, Gonzalez A, Gafni A, Tonmyr L, Barr R, Marcellus L, Varcoe C, Waddell C. Effects of nurse-home visiting on intimate partner violence and maternal income, mental health and self-efficacy by 24 months postpartum: a randomised controlled trial (British Columbia Healthy Connections Project). BMJ Open. 2025 Jan 6;15(1):e083147. doi: 10.1136/bmjopen-2023-083147. PMID 39762105
- [Derived] Catherine NLA, MacMillan H, Cullen A, Zheng Y, Xie H, Boyle M, Sheehan D, Lever R, Jack SM, Gonzalez A, Gafni A, Tonmyr L, Barr R, Marcellus L, Varcoe C, Waddell C. Effectiveness of nurse-home visiting in improving child and maternal outcomes prenatally to age two years: a randomised controlled trial (British Columbia Healthy Connections Project). J Child Psychol Psychiatry. 2024 May;65(5):644-655. doi: 10.1111/jcpp.13846. Epub 2023 Jul 19. PMID 37464862
- [Derived] Catherine NLA, Boyle M, Zheng Y, McCandless L, Xie H, Lever R, Sheehan D, Gonzalez A, Jack SM, Gafni A, Tonmyr L, Marcellus L, Varcoe C, Cullen A, Hjertaas K, Riebe C, Rikert N, Sunthoram A, Barr R, MacMillan H, Waddell C. Nurse home visiting and prenatal substance use in a socioeconomically disadvantaged population in British Columbia: analysis of prenatal secondary outcomes in an ongoing randomized controlled trial. CMAJ Open. 2020 Oct 27;8(4):E667-E675. doi: 10.9778/cmajo.20200063. Print 2020 Oct-Dec. PMID 33109532
- [Derived] Catherine NLA, Lever R, Marcellus L, Tallon C, Sheehan D, MacMillan H, Gonzalez A, Jack SM, Waddell C. Retaining participants in community-based health research: a case example on standardized planning and reporting. Trials. 2020 May 11;21(1):393. doi: 10.1186/s13063-020-04328-9. PMID 32393334
- [Derived] Catherine NLA, Lever R, Sheehan D, Zheng Y, Boyle MH, McCandless L, Gafni A, Gonzalez A, Jack SM, Tonmyr L, Varcoe C, MacMillan HL, Waddell C; British Columbia Healthy Connections Project Scientific Team. The British Columbia Healthy Connections Project: findings on socioeconomic disadvantage in early pregnancy. BMC Public Health. 2019 Aug 22;19(1):1161. doi: 10.1186/s12889-019-7479-5. PMID 31438906
- [Derived] Gonzalez A, Catherine N, Boyle M, Jack SM, Atkinson L, Kobor M, Sheehan D, Tonmyr L, Waddell C, MacMillan HL; Healthy Foundations Study Team. Healthy Foundations Study: a randomised controlled trial to evaluate biological embedding of early-life experiences. BMJ Open. 2018 Jan 26;8(1):e018915. doi: 10.1136/bmjopen-2017-018915. PMID 29374668
- [Derived] Catherine NL, Gonzalez A, Boyle M, Sheehan D, Jack SM, Hougham KA, McCandless L, MacMillan HL, Waddell C; British Columbia Healthy Connections Project Scientific Team. Improving children's health and development in British Columbia through nurse home visiting: a randomized controlled trial protocol. BMC Health Serv Res. 2016 Aug 4;16(a):349. doi: 10.1186/s12913-016-1594-0. PMID 27488474
- See also: Related Info — http://childhealthpolicy.ca/bc-healthy-connections-project/